CLINICAL TRIAL: NCT01514201
Title: A Phase I/II Study of ABT-888, An Oral Poly(ADP-ribose) Polymerase Inhibitor, and Concurrent Radiation Therapy, Followed by ABT-888 and Temozolomide, in Children With Newly Diagnosed Diffuse Pontine Gliomas (DIPG)
Brief Title: Veliparib, Radiation Therapy, and Temozolomide in Treating Younger Patients With Newly Diagnosed Diffuse Pontine Gliomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00082; NCI-2012-00082 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-033; 12-C-0213; CDR0000717423; P12978; PBTC-033 (Other: Pediatric Brain Tumor Consortium); PBTC-033 (Other: CTEP); U01CA081457 (NIH); UM1CA081457 (NIH); NCT01507324 (obsolete NCT alias)
Record Dates: First submitted 2012-01-16; First posted 2012-01-23 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Anaplastic Astrocytoma; Brain Stem Glioma; Childhood Mixed Glioma; Fibrillary Astrocytoma; Giant Cell Glioblastoma; Glioblastoma; Gliosarcoma; Untreated Childhood Anaplastic Astrocytoma; Untreated Childhood Brain Stem Glioma; Untreated Childhood Fibrillary Astrocytoma; Untreated Childhood Giant Cell Glioblastoma; Untreated Childhood Glioblastoma; Untreated Childhood Gliosarcoma
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Gliosarcoma | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Temozolomide; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (veliparib, temozolomide, 3D-CRT, IMRT) (Experimental): DOSE-ESCALATION: Patients receive veliparib PO BID 5 days a week for 6-7 weeks. Patients also undergo concurrent 3D-CRT or IMRT QD 5 days a week for 6-7 weeks.
  MAINTENANCE THERAPY: Beginning 3-4 weeks later, patients receive veliparib PO BID on days 1-5 and temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temozolomide; Drug: Veliparib

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D-CRT
  Other Names: 3-dimensional radiation therapy; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Optional correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I/II trial studies the side effects and the best dose of veliparib when given together with radiation therapy and temozolomide and to see how well they work in treating younger patients newly diagnosed with diffuse pontine gliomas. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells either by killing the cells or by stopping them from dividing. Giving veliparib with radiation therapy and temozolomide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the maximum-tolerated dose or recommended Phase II dose of ABT-888 (veliparib) which can be safely administered concurrently with radiation therapy, followed by maintenance therapy with ABT-888 and temozolomide (TMZ), in patients with newly diagnosed diffuse pontine gliomas (DIPG). (Phase I) II. To study the plasma pharmacokinetics (PK) of ABT-888 during ABT-888 and radiation therapy. (Phase I) III. To study the feasibility of intra-patient dose escalation of TMZ during maintenance therapy with ABT-888 and TMZ. (Phase I) IV. To describe the toxicities associated with administering ABT-888 and radiation therapy, followed by ABT-888 and TMZ, in patients with newly diagnosed DIPG. (Phase I) V. To estimate the proportion of newly diagnosed DIPG patients treated on protocol that are determined to have experienced pseudo progression. (Phase I) VI. To estimate the overall survival distribution for newly diagnosed patients with DIPG treated with the combination of ABT-888 and radiation therapy, followed by ABT-888 and TMZ, and compare to Pediatric Brain Tumor Consortium (PBTC) historical controls. (Phase II) VII. To study the feasibility of intra-patient dose escalation of TMZ during maintenance therapy with ABT-888 and TMZ. (Phase II) VIII. To estimate the proportion of newly diagnosed DIPG patients treated on protocol that are determined to have experienced pseudo progression. (Phase II)

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival (PFS) distribution and to summarize the best tumor responses observed prior to progression or recurrence.

II. To explore the plasma PK of ABT-888 during ABT-888 and radiation therapy. III. To explore peripheral blood mononuclear cell (PBMC) poly (ADP-ribose) polymerase 1(PARP) activity before and after treatment with ABT-888.

IV. To explore quantifying non-homologous end-joining (NHEJ) activity or gamma-H2A histone family, member X (H2AX) levels (as surrogate markers of unrepaired double-strand breaks (DSBs)) in PBMC before and after treatment with ABT-888.

V. To explore quantifying PARP activity and deoxyribonucleic acid (DNA)-repair protein levels in biopsied atypical pontine gliomas, if available.

VI. To explore associations of molecular parameters from secondary aims III, IV, and V with PFS and overall survival (OS) after conclusion of clinical trial.

VII. To explore the quantitative magnetic resonance (MR) measures of relative cerebral blood volume (rCBV), vascular permeability (Ktrans, fractional plasma volume [vp], and extravascular extracellular space volume fraction [ve] values), and apparent diffusion coefficient (ADC) within the first six months of initiating protocol treatment to correlate with disease outcome and determine whether such metrics differentiate patients with pseudo progression from those with true early progressive disease.

VIII. To explore the potential utility of urine biomarkers as a novel, non-invasive method of detecting and tracking changes in the status of pediatric brain stem gliomas.

OUTLINE: This is a phase I, dose-escalation study of veliparib followed by a phase II study.

DOSE-ESCALATION: Patients receive veliparib orally (PO) twice daily (BID) 5 days a week for 6-7 weeks. Patients also undergo concurrent 3-dimensional conformal radiotherapy (3D-CRT) or intensity-modulated radiotherapy (IMRT) once daily (QD) 5 days a week for 6-7 weeks.

MAINTENANCE THERAPY: Beginning 3-4 weeks later, patients receive veliparib PO BID on days 1-5 and temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed diffuse intrinsic pontine gliomas (DIPGs), defined as tumors with a pontine epicenter and diffuse intrinsic involvement of the pons, are eligible without histologic confirmation; patients with brainstem tumors that do not meet these criteria or not considered to be typical intrinsic pontine gliomas will only be eligible if the tumors are biopsied and proven to be an anaplastic astrocytoma, glioblastoma multiforme, gliosarcoma, anaplastic mixed glioma, or fibrillary astrocytoma

  * Patients with juvenile pilocytic astrocytoma, pilomyxoid astrocytoma, fibrillary astrocytoma, gangliogliomas, or other mixed gliomas without anaplasia are not eligible;
  * Patients with disseminated disease are not eligible, and magnetic resonance imaging (MRI) of spine must be performed if disseminated disease is suspected by the treating physician
* Patient must be able to swallow oral medications to be eligible for study enrollment
* Karnofsky >= 50% for patients > 16 years of age or Lansky >= 50% for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have not received any prior therapy other than surgery and/or steroids
* Absolute neutrophil count >= 1,000/mm^3
* Platelets >= 100,000/mm^3 (unsupported)
* Hemoglobin >= 10 g/dL (unsupported)
* Total bilirubin =< 1.5 times upper limit of normal (ULN) for age
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 5 x institutional upper limit of normal for age
* Albumin >= 2 g/dL
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 0.6 mg/dL (1 to < 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (>= 16 years of age)
* Female patients of childbearing potential must not be pregnant or breast-feeding; female patients of childbearing potential must have a negative serum or urine pregnancy test
* Patients of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study
* Signed informed consent according to institutional guidelines must be obtained; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that would compromise the patient's ability to tolerate protocol therapy or would likely interfere with the study procedures or results
* Patients with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy
* Patients with active seizures or a history of seizure are not eligible for study entry, with the exception of patients with documented febrile seizure

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Baxter, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (12):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Pediatric Brain Tumor Consortium, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Sesen J, Driscoll J, Shah N, Moses-Gardner A, Luiselli G, Alexandrescu S, Zurakowski D, Baxter PA, Su JM, Pricola Fehnel K, Smith ER. Neogenin is highly expressed in diffuse intrinsic pontine glioma and influences tumor invasion. Brain Res. 2021 Jul 1;1762:147348. doi: 10.1016/j.brainres.2021.147348. Epub 2021 Feb 9. No abstract available. PMID 33571520
- [Derived] Baxter PA, Su JM, Onar-Thomas A, Billups CA, Li XN, Poussaint TY, Smith ER, Thompson P, Adesina A, Ansell P, Giranda V, Paulino A, Kilburn L, Quaddoumi I, Broniscer A, Blaney SM, Dunkel IJ, Fouladi M. A phase I/II study of veliparib (ABT-888) with radiation and temozolomide in newly diagnosed diffuse pontine glioma: a Pediatric Brain Tumor Consortium study. Neuro Oncol. 2020 Jun 9;22(6):875-885. doi: 10.1093/neuonc/noaa016. PMID 32009149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients up to 21 years of age with newly diagnosed diffuse intrinsic pontine gliomas (DIPGs) were enrolled at Pediatric Brain Tumor Consortium (PBTC) member institutions. The first patient was enrolled on 2/1/2012 and the last patient was enrolled on 01/20/2016.
Pre-assignment Details: Of the 66 patients enrolled, 1 phase II patient was deemed ineligible due to an elevated alanine aminotransferase (ALT). Of note, the 6 phase I patients who were treated at the established maximum tolerated dose (MTD) during the phase I portion of the trial were also counted as phase II patients in analyses of phase II objectives.
Groups:
- Phase I, Dose Level 1 (50 mg); Phase I, Dose Level 2 (65 mg); Phase I, Dose Level 3 (85 mg): Dose Escalation: Patients receive veliparib orally (PO) twice a day (BID) 5 days a week for 6-7 weeks. Patients also undergo concurrent 3-dimensional conformal radiation therapy (3D-CRT) or intensity modulated radiation therapy (IMRT) once a day (QD) 5 days a week for 6-7 weeks.
  Maintenance Therapy: Beginning 3-4 weeks later, patients receive veliparib PO BID on days 1-5 and temozolomide (TMZ) PO QD on days 1-5. Treatment repeats every 28 days for up to 10 courses in the absence of disease progression or unacceptable toxicity. All patients start maintenance with 25 mg/m2 BID of veliparib and 135 mg/m2/day of TMZ. Intra-patient escalation of TMZ to 175 mg/m2/day and 200 mg/m2/day in subsequent courses was allowed for patients with minimal toxicities. However this intra-patient dose escalation was halted early as it was not well tolerated.
- Phase II (MTD): Patients receive veliparib at the maximum tolerated dose (MTD) orally (PO) twice a day (BID) 5 days a week for 6-7 weeks. Patients also undergo 3-dimensional conformal radiation therapy (3D-CRT) or intensity modulated radiation therapy (IMRT) once a day (QD) 5 days a week for 6-7 weeks.
  Maintenance Therapy: Beginning 3-4 weeks later, patients receive veliparib PO BID on days 1-5 and temozolomide (TMZ) PO QD on days 1-5. Treatment repeats every 28 days for up to 10 courses in the absence of disease progression or unacceptable toxicity. All patients start maintenance with 25 mg/m2 BID of veliparib and 135 mg/m2/day of TMZ. Intra-patient escalation of TMZ to 175 mg/m2/day and 200 mg/m2/day in subsequent courses was allowed for patients with minimal toxicities. However this intra-patient dose escalation was halted early (before the phase II study was initiated) as it was not well tolerated.
Period: PHASE I: Veliparib + Radiation Therapy
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Started | 6 | 6 | 6 | 0
Completed | 5 | 6 | 6 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Period: PHASE I: Maintenance With Veliparib/TMZ
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Started | 5 | 6 | 6 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 5 | 6 | 6 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 4 | 4 | 5 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Period: PHASE II: Veliparib + Radiation Therapy
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Started | 0 | 0 | 0 | 47
Completed | 0 | 0 | 0 | 35
Not Completed | 0 | 0 | 0 | 12
Not completed — Ineligible | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 6
Period: PHASE II: Maintenance With Veliparib/TMZ
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Started | 0 | 0 | 0 | 35
Completed | 0 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 33
Not completed — Adverse Event | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 7
Not completed — Lack of Efficacy | 0 | 0 | 0 | 22

BASELINE CHARACTERISTICS:
Population: The one ineligible patient enrolled on the protocol was excluded. Summary statistics for baseline characteristics are shown for eligible patients only (n=65).
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 47 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 6 | 47 | 65
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 6.3 [5.3 to 10.4] | 10.2 [5.4 to 12.9] | 9.2 [2.2 to 15.8] | 6.5 [2.5 to 11.6] | 6.6 [2.2 to 15.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 30 | 37
  Male | 4 | 3 | 4 | 17 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 7 | 10
  Not Hispanic or Latino | 3 | 5 | 5 | 34 | 47
  Unknown or Not Reported | 0 | 1 | 1 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 2
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 2 | 1 | 9 | 12
  White | 3 | 3 | 5 | 29 | 40
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 6 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 6 | 47 | 65

OUTCOME MEASURES:

1. Primary Outcome: Maximum-tolerated Dose of Veliparib Defined as Highest Dose Level With Fewer Than 2 Dose Limiting Toxicities in 6 Patients as Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (Phase I)
Description: The traditional 3+3 dose finding algorithm was used to estimate the maximum-tolerated dose of veliparib given concurrently with radiation therapy. The dose-limiting toxicity observation period was the first 10 weeks of therapy. Dose-limiting toxicities included any grade 4 non-hematologic toxicity, any grade 3 non-hematologic toxicity with a few exceptions (see section 5.2.1.2 of the protocol document), any grade 2 non-hematologic toxicity that persisted for >7 days and considered medically significant that required treatment interruption; grade 3 or higher thrombocytopenia or grade 4 neutropenia; and any Veliparib related adverse event that led to a dose reduction or the permanent cessation of therapy.
Time Frame: 10 weeks
Population: The first 18 patients enrolled on the study were phase I patients used to determine the maximum tolerated dose or the recommended phase II dose and to address other objectives of the phase I component of this trial.
Measure: Number; unit: mg/m2/dose BID
Groups:
- Phase I Patients: The first 18 patients enrolled on the study were phase I patients used to determine the maximum tolerated dose or the recommended phase II dose and to address other objectives of the phase I component of this trial. The starting dose level was 50 mg/m2/dose twice a day (BID) and other dose levels to be studied were 65 and 85 mg/m2/dose BID. If the 85 mg/m2 dose level was tolerated, there was a plan to study a higher dose level (110 mg/m2/dose BID) but only if supported by clinical data.
Arm/Group | Phase I Patients
Number analyzed (Participants) | 18
mg/m2/dose BID | 65

2. Primary Outcome: Percentage of Participants Observed to Have Unacceptable Toxicity During the Intra-patient Dose Escalation of Temozolomide During Maintenance Therapy (Feasibility Analysis Population)
Description: Unacceptable toxicities during maintenance included events at least possibly attributable to Veliparib and temozolomide (TMZ) such as any grade 4 non-hematologic toxicity, any grade 3 non-hematologic toxicity with some exceptions (e.g., grade 3 nausea/vomiting <5 days, grade 3 fever or infection <5 days), grade 3+ thrombocytopenia, grade 4 neutropenia, delay >14 days in starting subsequent cycle due to neutrophil <1,000/mm3 or platelet <100,000/mm3. Maintenance therapy was initiated with 25 mg/m2 Veliparib and 135 mg/m2 of TMZ, with the possibility to escalate TMZ to 175 mg/m2 and 200 mg/m2 in courses 2 and 3, respectively, if no unacceptable toxicities occurred following one course of treatment at each of the dose levels to be tested. Intra-patient dose escalation to a given dose (135, 175, or 200 mg/m2) was halted based on rules employed in 3+3 designs. This dose escalation was intended for all patients but was halted early, during the phase I portion, as it was not well tolerated.
Time Frame: 28 days per treatment cycle
Population: Patients were combined across dose levels since they received the same maintenance therapy. Though this objective was intended for all patients, only the first 12 enrolled were included as the dose-escalation stopped early. 1 of the first 12 patients did not start maintenance due to early progression, so 11 patients started dose level 1.
Measure: Number; unit: % of participants
Groups:
- Dose Level 1 (135 mg/m2): Participants in the feasibility analysis population that started dose level 1 of the intra-patient dose escalation during maintenance (Veliparib 25 mg/m2 twice a day (BID) + temozolomide 135 mg/m2/day)
- Dose Level 2 (175 mg/m2): Participants in the feasibility analysis population that started dose level 2 of the intra-patient dose escalation during maintenance (Veliparib 25 mg/m2 twice a day (BID) + temozolomide 175 mg/m2/day)
- Dose Level 3 (200 mg/m2): Participants in the feasibility analysis population that started dose level 1 of the intra-patient dose escalation during maintenance (Veliparib 25 mg/m2 twice a day (BID) + temozolomide 200 mg/m2/day)
Arm/Group | Dose Level 1 (135 mg/m2) | Dose Level 2 (175 mg/m2) | Dose Level 3 (200 mg/m2)
Number analyzed (Participants) | 11 | 5 | 3
% of participants | 9 | 40 | 67
Statistical Analysis 1: Comparison: Dose Level 1 (135 mg/m2) vs Dose Level 2 (175 mg/m2) vs Dose Level 3 (200 mg/m2); Intra-patient dose escalation of temozolomide during maintenance was assessed based on similar rules employed in traditional 3+3 designs. For example intra-patient dose escalation would be halted if at any time 2 out of first 2-6 patients experienced dose-modifying toxicities at a given dose level or if 4 out of first 12 patients experienced dose-modifying toxicities at a given dose level; Test type: Other — This was descriptive in nature. Two of the first 5 patients who were escalated to 175 mg/m2 of temozolomide during the maintenance intra-patient dose escalation had dose-modifying toxicities (DMTs). Since the ad hoc stopping rule was met, intra-patient dose escalation was halted and all subsequent patients were to receive 135 mg/m2 of temozolomide during maintenance; Percentage of patients with DMTs = 40

3. Primary Outcome: Overall Survival
Description: Overall survival was defined as the interval from date on treatment to date of death from any cause or to date of last follow-up. Patients who had not failed (died) at the time of analyses were censored at their last date of contact. The method of Kaplan and Meier was used to estimate overall survival. The 3-year estimate with a 95% confidence interval is reported.
Time Frame: Time from initiation of therapy to the date of death from any cause or to the date patient was known to be alive for surviving patients, assessed to up to 3 years
Population: 53 patients were evaluable for outcome analyses (47 phase II patients + 6 phase I patients treated at the MTD). 50 patients were evaluable; 1 patient withdrew prior to beginning protocol therapy and 2 patients did not receive adequate study drug to be evaluable for efficacy. To be evaluable patients had to receive at least one dose of Veliparib.
Measure: Number (95% Confidence Interval); unit: Percent probability
Groups:
- Phase II Patients + Phase I MTD Patients: Phase II patients were those enrolled after the maximum tolerated dose was established in the phase I portion of this trial. Six patients enrolled as phase I patients but who were treated with the established maximum tolerated dose of 65 mg/m2/day twice a day (BID) were also considered phase II patients. There were 53 eligible phase II patients (including the latter six patients). Fifty (50) of these patients were evaluable for outcome analyses as 1 patient withdrew prior to beginning protocol therapy and 2 other patients did not receive adequate study drug to be evaluable for efficacy. To be evaluable for assessing overall survival, patients had to receive at least one dose of Veliparib.
Arm/Group | Phase II Patients + Phase I MTD Patients
Number analyzed (Participants) | 50
Percent probability | 5.3 [0.0 to 12.4]

4. Primary Outcome: Number of Phase I Patients Who Experienced Dose Limiting Toxicities (DLTs)
Description: DLTs were defined as any of the following adverse events that were at least possibly attributable to Veliparib observed during the dose finding phase (the first 10 weeks of therapy). Hematologic dose limiting toxicities included grade 3 and higher thrombocytopenia or grade 4 neutropenia. Non-hematologic dose limiting toxicities included any grade 4 non-hematologic toxicity, any grade 3 non-hematologic toxicity with some exceptions (e.g., nausea and vomiting of <5 days; fever or infection of <5 days; hypophosphatemia, hypokalemia, hypocalcemia or hypomagnesemia responsive to oral supplementation; elevation of transaminases that return to levels meeting eligibility criteria within 7 days), or any grade non-hematologic toxicity that persisted for >7 days and considered medically significant or sufficiently intolerable by patients that required treatment interruption.
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg)
Number analyzed (Participants) | 6 | 6 | 6
Participants | 1 | 0 | 3

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the interval from date of treatment initiation to date of first event (disease progression or relapse, second malignancy or death from any cause). Patients who had not failed at the time of analyses were censored at their last date of contact. The method of Kaplan and Meier was used to estimate PFS. A 3-year estimate with a 95% confidence interval is reported.
Time Frame: Time from initiation of treatment to the earliest date of failure (disease progression, death from any cause, or second malignancy), assessed up to 3 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percent probability
Groups:
- Phase II Patients + Phase I MTD Patients: Phase II patients were those enrolled after the maximum tolerated dose was established in the phase I portion of this trial. Six patients enrolled as phase I patients but who were treated with the established maximum tolerated dose of 65 mg/m2/day twice a day (BID) were also considered phase II patients. There were 53 eligible phase II patients (including the latter six patients). Fifty (50) of these patients were evaluable for outcome analyses as 1 patient withdrew prior to beginning protocol therapy and 2 other patients did not receive adequate study drug to be evaluable for efficacy. To be evaluable for assessing PFS, patients had to receive at least one dose of Veliparib.
Arm/Group | Phase II Patients + Phase I MTD Patients
Number analyzed (Participants) | 50
Percent probability | 2.9 [0.0 to 6.8]

6. Secondary Outcome: Percentage of Patients With Pseudo Progression
Description: For participants that showed possible tumor progression (pseudo progression) on magnetic resonance imaging (MRI) during the first 6 months of therapy, treating physicians had the option of allowing patients to remain on therapy and repeating the disease assessment in 4-6 weeks. If the repeat MRI at 4-6 weeks showed disease progression, the patient was noted to have true disease progression (and the progression date corresponded to that of the first MRI). If the repeat MRI at 4-6 weeks did not show disease progression, then the patient was noted to have pseudo progression. The percentage of patients observed to have experienced pseudo progression was provided with a 95% confidence interval.
Time Frame: Up to 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Number analyzed (Participants) | 6 | 6 | 6 | 47
Percentage of participants | 33.3 [6.3 to 72.9] | 16.7 [0.9 to 59.8] | 0 [0.0 to 40.2] | 12.8 [5.7 to 24.5]

7. Secondary Outcome: Maximum Concentration of Veliparib (Cmax) on Days 1 and 4 (Measured in ng/mL) [Pharmacokinetic Parameter]
Description: During course 1, blood samples were collected pre-veliparib on day 1, at 0.5, 1, 2, and 6-8 hours after the first dose, pre-veliparib on day 4 (steady state), and 2 hours after the morning dose. Veliparib concentrations were measured using a liquid chromatography tandem mass spectrometry assay and pharmacokinetic parameters were evaluated using a non-compartmental analysis. Cmax measures the highest concentration of drug.
Time Frame: Up to day 4
Population: Pharmacokinetic studies were optional for the phase II portion of the study. Pharmacokinetic data were not available for all patients as indicated in the outcome measure data table below.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Number analyzed (Participants) | 6 | 6 | 6 | 47
ng/mL
  Day 1, Cmax (ng/mL): number analyzed (Participants) | 6 | 6 | 4 | 25
  Day 1, Cmax (ng/mL) | 519 (241) | 843 (364) | 1074 (372) | 844 (279)
  Day 4, Cmax (ng/mL): number analyzed (Participants) | 6 | 6 | 4 | 19
  Day 4, Cmax (ng/mL) | 409 (84) | 788 (435) | 954 (348) | 717 (232)

8. Secondary Outcome: Mean Apparent Clearance (CL/F) for Veliparib [Pharmacokinetic Parameter]
Description: During course 1, blood samples were collected pre-veliparib on day 1, at 0.5, 1, 2, and 6-8 hours after the first dose, pre-veliparib on day 4 (steady state), and 2 hours after the morning dose. Veliparib concentrations were measured using a liquid chromatography tandem mass spectrometry assay and pharmacokinetic parameters were evaluated using a non-compartmental analysis.
Time Frame: Up to day 4
Population: Pharmacokinetic studies were optional for the phase II portion of the study. 6/6 phase I dose level 1 patients, 6/6 phase I dose level 2 patients, 4/6 phase I dose level 3 patients, and 25/47 phase II patients had this data available.
Measure: Mean (Standard Deviation); unit: L/m^2/h
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Number analyzed (Participants) | 6 | 6 | 4 | 25
L/m^2/h | 16.1 (8.1) | 13.2 (4.3) | 15.8 (8.3) | 11.7 (8.8)

9. Secondary Outcome: Maximum Concentration of Veliparib (Cmax) on Day 1 (Measured in μM) [Pharmacokinetic Parameter]
Description: as for outcome 7
Time Frame: Day 1
Population: Pharmacokinetic studies were optional for the phase II portion of the study. Pharmacokinetic data were not available for all patients. 6/6 phase I dose level 1, 6/6 phase I dose level 2, 4/6 phase I dose level 3, and 25/47 phase II patients had day 4 Cmax data available.
Measure: Mean (Standard Deviation); unit: μM
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Number analyzed (Participants) | 6 | 6 | 4 | 25
μM | 2.12 (0.98) | 3.45 (1.49) | 4.40 (1.52) | 3.45 (1.14)

10. Other Pre Specified Outcome: Percentage of Participants With Significant Changes in Poly(ADP-ribose) Polymerase (PARP) Levels Post-Veliparib, as Measured in Peripheral Blood Monocytes (PBMCs)
Description: Blood samples were collected from patients and assessed pre- and post-Veliparib to assess treatment-induced changes. A significant change in PBMC PARP level was arbitrarily defined as a >50% increase or decrease from the pre-treatment level, documented at week 6 and/or week 11 after starting protocol therapy.
Time Frame: Baseline and up to 11 weeks
Population: Only 27 patients had pre- and post-Veliparib samples available in order to assess treatment-related changes. Two of the patients had inconsistent changes in post-Veliparib PARP levels and therefore were excluded from the analysis, leaving 25 patients for this objective.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase I, Dose Level 1 (50 mg); Phase I, Dose Level 2 (65 mg); Phase I, Dose Level 3 (85 mg): Dose Escalation: Patients receive veliparib orally (PO) twice a day (BID) 5 days a week for 6-7 weeks. Patients also undergo concurrent 3D conformal radiation therapy (3D-CRT) or intensity modulated radiation therapy (IMRT) once a day (QD) 5 days a week for 6-7 weeks.
  Maintenance Therapy: Beginning 3-4 weeks later, patients receive veliparib PO BID on days 1-5 and temozolomide (TMZ) PO QD on days 1-5. Treatment repeats every 28 days for up to 10 courses in the absence of disease progression or unacceptable toxicity. All patients start maintenance with 25 mg/m2 BID of veliparib and 135 mg/m2/day of TMZ. Intra-patient escalation of TMZ to 175 mg/m2/day and 200 mg/m2/day in subsequent courses was allowed for patients with minimal toxicities. However this intra-patient dose escalation was halted early as it was not well tolerated.
- Phase II (MTD): Patients receive veliparib at the maximum tolerated dose (MTD) orally (PO) twice a day (BID) 5 days a week for 6-7 weeks. Patients also undergo 3D conformal radiation therapy (3D-CRT) or intensity modulated radiation therapy (IMRT) once a day (QD) 5 days a week for 6-7 weeks.
  Maintenance Therapy: Beginning 3-4 weeks later, patients receive veliparib PO BID on days 1-5 and temozolomide (TMZ) PO QD on days 1-5. Treatment repeats every 28 days for up to 10 courses in the absence of disease progression or unacceptable toxicity. All patients start maintenance with 25 mg/m2 BID of veliparib and 135 mg/m2/day of TMZ. Intra-patient escalation of TMZ to 175 mg/m2/day and 200 mg/m2/day in subsequent courses was allowed for patients with minimal toxicities. However this intra-patient dose escalation was halted early (before the phase II study was initiated) as it was not well tolerated.
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Number analyzed (Participants) | 3 | 4 | 4 | 14
percentage of participants | 100 [37 to 100] | 100 [47 to 100] | 75 [25 to 99] | 36 [15 to 63]

11. Other Pre Specified Outcome: Change in Non-homologous End-joining (NHEJ) Activity as Measured in Peripheral Blood Monocytes (PBMCs)
Description: Levels of non-homologous end-joining (NHEJ) activity were to be calculated. Cox models to explore associations between the levels of NHEJ and outcome (progression-free survival and overall survival) were planned, in addition to looking at associations between Poly(ADP-ribose) polymerase (PARP) activity and NHEJ levels.
Time Frame: Baseline to up to 3 years
Population: These data were not available as the lab did not perform these analyses. There are no plans to perform these analyses.
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Other Pre Specified Outcome: Change in Level of Gamma-H2A Histone Family, Member X (H2AX) Measured in PBMCs
Description: Levels of gamma-H2A histone family, member X (H2AX) were to be calculated. Cox models to explore associations between the levels of gamma-H2AX and outcome (progression-free survival and overall survival) were planned, in addition to looking at associations between Poly(ADP-ribose) polymerase (PARP) activity and gamma-H2AX levels.
Time Frame: Baseline to up to 3 years
Population: These data were not available as the lab did not perform these analyses. There are no plans to perform these analyses.
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Other Pre Specified Outcome: Levels of Urinary Biomarkers
Description: Urine samples were analyzed for a panel of biomarkers. Netrin-1 levels were determined by ELISA. Levels of matrix metalloproteinase 3 (MMP3) and basic fibroblast growth factor (bFGF) were analyzed using custom Luminex® screening assays. Tissue inhibitor of metalloproteinase 1 (TIMP1) levels were analyzed using a Luminex® performance assay. Protein concentrations are given in picograms per microgram (pg/μg), and were determined by dividing the concentration of the target protein in the sample (pg/mL) by the concentration of total protein in the sample (μg/mL) as a normalization measure.
Time Frame: Baseline to up to 3 years
Population: Not all patients had urine samples at each time point.
Measure: Median (Full Range); unit: pg/μg
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Number analyzed (Participants) | 6 | 6 | 6 | 47
pg/μg
  MMP3 at pre-study: number analyzed (Participants) | 5 | 6 | 3 | 35
  MMP3 at pre-study | 2.0 [0.9 to 3.2] | 1.0 [0.4 to 2.1] | 0.0 [0.0 to 2.6] | 1.1 [0.0 to 7.6]
  MMP3 at week 10-11: number analyzed (Participants) | 5 | 5 | 5 | 24
  MMP3 at week 10-11 | 1.4 [0.7 to 4.0] | 1.0 [0.0 to 2.9] | 0.8 [0.4 to 3.5] | 2.6 [0.0 to 9.8]
  MMP3 at week 18: number analyzed (Participants) | 3 | 3 | 3 | 18
  MMP3 at week 18 | 4.3 [4.2 to 4.6] | 1.7 [1.3 to 2.4] | 0.7 [0.5 to 1.0] | 2.3 [0.0 to 15.8]
  MMP3 at week 26: number analyzed (Participants) | 2 | 2 | 2 | 11
  MMP3 at week 26 | 2.9 [2.8 to 3.0] | 0.4 [0.3 to 0.5] | 1.0 [1.0 to 1.1] | 3.0 [0.2 to 6.4]
  Netrin-1 at pre-study: number analyzed (Participants) | 5 | 6 | 3 | 35
  Netrin-1 at pre-study | 0.1 [0.0 to 0.3] | 0.1 [0.1 to 0.2] | 0.1 [0.0 to 0.3] | 0.1 [0.0 to 0.9]
  Netrin-1 at week 10-11: number analyzed (Participants) | 5 | 4 | 4 | 24
  Netrin-1 at week 10-11 | 0.1 [0.1 to 0.3] | 0.1 [0.0 to 0.3] | 0.1 [0.0 to 0.5] | 0.0 [0.0 to 0.3]
  Netrin-1 at week 18: number analyzed (Participants) | 3 | 2 | 3 | 18
  Netrin-1 at week 18 | 0.3 [0.2 to 0.3] | 0.1 [0.1 to 0.1] | 0.0 [0.0 to 0.0] | 0.1 [0.0 to 0.6]
  Netrin-1 at week 26: number analyzed (Participants) | 2 | 2 | 1 | 11
  Netrin-1 at week 26 | 0.4 [0.4 to 0.4] | 0.2 [0.2 to 0.3] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 1.0]
  TIMP1 at pre-study: number analyzed (Participants) | 5 | 6 | 3 | 35
  TIMP1 at pre-study | 3.4 [3.1 to 9.0] | 9.9 [1.4 to 18.7] | 10.8 [1.5 to 39.7] | 7.3 [1.9 to 16.8]
  TIMP1 at week 10-11: number analyzed (Participants) | 5 | 6 | 5 | 24
  TIMP1 at week 10-11 | 6.2 [4.0 to 22.4] | 11.9 [0.0 to 40.5] | 12.3 [7.8 to 143.7] | 7.5 [3.5 to 20.3]
  TIMP1 at week 18: number analyzed (Participants) | 3 | 3 | 3 | 18
  TIMP1 at week 18 | 10.7 [2.9 to 18.1] | 7.7 [5.8 to 9.6] | 14.8 [12.0 to 61.9] | 7.1 [2.4 to 44.7]
  TIMP1 at week 26: number analyzed (Participants) | 2 | 2 | 2 | 11
  TIMP1 at week 26 | 7.3 [7.2 to 7.4] | 5.2 [2.6 to 7.8] | 32.8 [4.9 to 60.7] | 10.7 [2.4 to 30.8]
  bFGF at pre-study: number analyzed (Participants) | 5 | 6 | 3 | 35
  bFGF at pre-study | 3.1 [1.3 to 7.8] | 1.9 [1.0 to 3.7] | 1.2 [0.0 to 3.0] | 4.5 [0.0 to 18.5]
  bFGF at week 10-11: number analyzed (Participants) | 5 | 5 | 5 | 24
  bFGF at week 10-11 | 3.6 [3.3 to 9.3] | 2.1 [0.8 to 6.4] | 1.8 [0.8 to 2.7] | 3.5 [0.0 to 9.4]
  bFGF at week 18: number analyzed (Participants) | 3 | 3 | 3 | 18
  bFGF at week 18 | 10.3 [7.1 to 10.9] | 3.5 [1.5 to 5.2] | 1.3 [0.6 to 1.4] | 4.4 [0.0 to 40.8]
  bFGF at week 26: number analyzed (Participants) | 2 | 2 | 2 | 11
  bFGF at week 26 | 7.7 [7.0 to 8.4] | 0.9 [0.6 to 1.2] | 1.1 [1.1 to 1.1] | 4.5 [0.3 to 66.0]

14. Secondary Outcome: Apparent Volume of Distribution (Vd/F) for Veliparib [Pharmacokinetic Parameter]
Description: as for outcome 8
Time Frame: Up to day 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L/m^2
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Number analyzed (Participants) | 6 | 6 | 4 | 25
L/m^2 | 75.4 (29.2) | 56.1 (25.4) | 63.9 (10.6) | 73.1 (109.7)

15. Secondary Outcome: Terminal Half-life (t1/2) for Veliparib [Pharmacokinetic Parameter]
Description: as for outcome 8
Time Frame: Up to day 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Number analyzed (Participants) | 6 | 6 | 4 | 25
Hour | 5.18 (6.34) | 2.62 (0.76) | 4.45 (4.80) | 2.18 (2.71)

16. Secondary Outcome: Trough for Veliparib [Pharmacokinetic Parameter]
Description: as for outcome 8
Time Frame: Up to day 4
Population: Pharmacokinetic studies were optional for the phase II portion of the study. 6/6 phase I dose level 1 patients, 5/6 phase I dose level 2 patients, 4/6 phase I dose level 3 patients, and 20/47 phase II patients had this data available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase I, Dose Level 1 (50 mg) | Phase I, Dose Level 2 (65 mg) | Phase I, Dose Level 3 (85 mg) | Phase II (MTD)
Number analyzed (Participants) | 6 | 5 | 4 | 20
ng/mL | 58 (19) | 140 (173) | 163 (97) | 84 (42)

ADVERSE EVENTS:
Time Frame: Approximately 1 year after starting treatment
Description: Adverse events (AEs) were graded according to CTCAE v4.0. AEs collected per protocol included: a) grade 1 and 2 AEs if attribution was at least possibly related to veliparib and b) all grade 3+ AEs on treatment and within 30 days off treatment. All AEs collected are reported. As the intra-patient escalation of TMZ during maintenance was by course (rather than patient) and was halted early (only 5(3) patients escalated to 175(200) mg/m2), AEs were not reported separately by course-specific doses.
Groups:
- Phase I, Dose Level 1 (50 mg/m2); Phase I, Dose Level 2 (65 mg/m2); Phase I, Dose Level 3 (85 mg/m2): Dose Escalation: Patients receive veliparib orally (PO) twice a day (BID) 5 days a week for 6-7 weeks. Patients also undergo concurrent radiation (3D-CRT or IMRT) once a day (QD) 5 days a week for 6-7 weeks.
  Maintenance Therapy: Beginning 3-4 weeks later, patients receive veliparib PO BID on days 1-5 and temozolomide (TMZ) PO QD on days 1-5. Treatment repeats every 28 days for up to 10 courses in the absence of disease progression or unacceptable toxicity. All patients start maintenance with 25 mg/m2 BID of veliparib and 135 mg/m2/day of TMZ. Intra-patient escalation of TMZ to 175 mg/m2/day and 200 mg/m2/day in subsequent courses was allowed for patients with minimal toxicities. However this intra-patient dose escalation was halted early as it was not well tolerated.
- Phase II (MTD): Patients receive veliparib at the maximum tolerated dose (MTD) orally (PO) twice a day (BID) 5 days a week for 6-7 weeks. Patients also undergo concurrent radiation (3D-CRT or IMRT) once a day (QD) 5 days a week for 6-7 weeks.
  Maintenance Therapy: Beginning 3-4 weeks later, patients receive veliparib PO BID on days 1-5 and temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 10 courses in the absence of disease progression or unacceptable toxicity. All patients start maintenance with 25 mg/m2 BID of veliparib and 135 mg/m2/day of TMZ. Intra-patient escalation of TMZ to 175 mg/m2/day and 200 mg/m2/day in subsequent courses was allowed for patients with minimal toxicities. However this intra-patient dose escalation was halted early (before the phase II study was initiated) as it was not well tolerated.
Arm/Group | Phase I, Dose Level 1 (50 mg/m2) | Phase I, Dose Level 2 (65 mg/m2) | Phase I, Dose Level 3 (85 mg/m2) | Phase II (MTD)
All-Cause Mortality (participants affected / at risk) | 6/6 | 5/6 | 6/6 | 40/47
Serious Adverse Events (participants affected / at risk) | 5/6 | 2/6 | 2/6 | 19/47
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 46/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Dose Level 1 (50 mg/m2) (N=6) | Phase I, Dose Level 2 (65 mg/m2) (N=6) | Phase I, Dose Level 3 (85 mg/m2) (N=6) | Phase II (MTD) (N=47)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 8 (9)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (3) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papilledema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Dose Level 1 (50 mg/m2) (N=6) | Phase I, Dose Level 2 (65 mg/m2) (N=6) | Phase I, Dose Level 3 (85 mg/m2) (N=6) | Phase II (MTD) (N=47)
Anemia (Blood and lymphatic system disorders) | 4 (11) | 4 (20) | 6 (13) | 27 (59)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (4) | 5 (6) | 1 (1) | 14 (19)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (7) | 5 (7) | 4 (7) | 14 (23)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (3) | 4 (11) | 4 (12) | 21 (35)
Fatigue (General disorders) | 4 (4) | 4 (5) | 3 (7) | 15 (26)
Fever (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (2) | 0 (0) | 23 (33)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 12 (22)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
GGT increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (11)
Lymphocyte count decreased (Investigations) | 5 (15) | 6 (34) | 6 (27) | 44 (260)
Neutrophil count decreased (Investigations) | 3 (8) | 4 (17) | 5 (24) | 19 (66)
Platelet count decreased (Investigations) | 5 (14) | 5 (30) | 4 (18) | 23 (72)
Weight gain (Investigations) | 2 (2) | 0 (0) | 0 (0) | 3 (4)
Weight loss (Investigations) | 0 (0) | 1 (1) | 2 (3) | 4 (4)
White blood cell decreased (Investigations) | 5 (17) | 5 (36) | 5 (22) | 36 (131)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 4 (4) | 10 (14)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (2) | 8 (11)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0) | 18 (33)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (6) | 2 (2) | 9 (21)
Hypokalemia (Metabolism and nutrition disorders) | 4 (8) | 0 (0) | 3 (4) | 14 (22)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (3) | 6 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 4 (5) | 14 (20)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (6)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Abducens nerve disorder (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 5 (5)
Ataxia (Nervous system disorders) | 4 (4) | 3 (4) | 1 (1) | 5 (9)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 3 (4) | 4 (5) | 7 (12)
IVth nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spasticity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 5 (6)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (5)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT01514201/Prot_SAP_000.pdf